CLINICAL TRIAL: NCT01335841
Title: Evaluation of an 3D Imaging Intensifier Coupled to a Navigation Station in the Surgery of the Spine and Pelvis
Acronym: FLUORONAV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AdministrateurCIC (Other)
Collaborators: PRAXIM company (Unknown)
Responsible Party: Sponsor-Investigator, AdministrateurCIC, principal investigator, University Hospital, Grenoble
Organization: University Hospital, Grenoble (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: DCIC-10 25
Record Dates: First submitted 2011-01-31; First posted 2011-04-14 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3D fluoroscopy and navigation station (Experimental)
  Interventions: Device: Navigation station coupled with a 3D fluoroscopy
- 2D and anatomical landmarks (Active Comparator)
  Interventions: Device: Navigation station coupled with a 3D fluoroscopy

INTERVENTIONS:
Device: Navigation station coupled with a 3D fluoroscopy — After randomization, patients will be operated with the conventional method either with navigation station. In the conventional method, the orthopedic surgeon based on anatomical criteria to establish its implants. It uses an image intensifier in 2D mode to monitor the implementation of the implants. In computer assisted surgery, the surgeon uses a navigation station that allows real-time flow instruments to guide its implementation of the implants. It uses an image intensifier in 3D mode on the one hand to achieve a first series of image that will be used for navigation and also to monitor the implementation of the implants.

SUMMARY:
The purpose of this study is to demonstrate an optimization of the establishment of orthopedic implants in surgery of the spine and pelvic ring by combining 3D fluoroscopy and navigation system versus conventional method involving anatomical landmarks and 2D fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years old
* Patient affiliated to social security or similarly regime
* Patient with a disease of the pelvic ring, with an indication of establishment of a screw sacro-iliac
* Patient with a disease of the spine, with an indication of establishment of pedicle implant

Exclusion Criteria:

* Intubated patient resuscitation
* Pregnant women and lactating mothers
* Adult unable to express their consent
* Ward of court or under guardianship
* Person under legal protection
* Person deprived of freedom by judicial or administrative decision
* Person hospitalized without their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Reading number of trips extra-pedicular or extra bone in both groups on a postoperative TDM | two years

SECONDARY OUTCOMES:
measure radiation of the surgeon and the patient in the two groups | two years
  delivered dose and irradiation time during the duration of the intervention for the sacro-iliac screw connections, or for the establishment of two pedicle screws in spinal surgery over a 2-D amplifier
Show that the operative time is not increased significantly taking into account the learning curve and the benefit provided from a conventional 2-D amplifier | two years
  comparison of operating times of interventions between "3D-navigation" and conventional methods

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Merloz, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Clinical Investigation Center - Technological Innovation - Inserm 803 - University Hospital France, Grenoble, France